CLINICAL TRIAL: NCT06611306
Title: BEAT-Breast - Improving Outcomes for Breast Cancer Patients With Brain Metastases: a Pilot Nonrandomised Single Arm Phase 2 Clinical Trial in Patients With Primary Breast Cancer With Brain Metastases Who Are Not Suitable for Stereotactic Radiotherapy
Brief Title: BEAT-Breast: Trial of DE-iPTV in Patients With Primary Breast Cancer With Brain Metastases Who Are Not Suitable for Stereotactic Radiotherapy.
Acronym: BEAT-Breast
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: University of Leicester (Other); Centro Nacional de Investigaciones Oncologicas CARLOS III (Other); East and North Hertfordshire NHS Trust (Other Government); Norfolk and Norwich University Hospitals NHS Foundation Trust (Other); Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C/46/2023
Record Dates: First submitted 2024-09-23; First posted 2024-09-24 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Brain Metastases, Adult; Breast Cancer
Keywords: Radiotherapy; Brain metastases; Metastatic Breast Cancer
MeSH Terms: conditions — Brain Neoplasms; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Non-randomised interventional multi-centre feasibility trial in patients with brain metastases from breast cancer receiving dose escalated internal PTV (DE-iPTV) radiotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DE-iPTV radiotherapy (Experimental): Patients will undergo a radiotherapy planning scan, and an upto date MRI brain with contrast. Patients will receive 5 fractions of DE-iPTV radiotherapy over 1 week.
  Interventions: Radiation: DE-iPTV

INTERVENTIONS:
Radiation: DE-iPTV — Dose-escalated VMAT-based radiotherapy, as previously described in our planning study

SUMMARY:
The aim of this study is to demonstrate if it is possible to delivering a novel and modern radiotherapy approach (Dose Escalated internal PTV (DE-iPTV)) and to collect health related quality of life in patients whose breast cancer has spread to the brain (brain metastases) at 8 weeks post enrolling into the study.

The main questions that have been set out to to answer are:

* Is it possible to deliver the novel radiotherapy approach, DE-iPTV?
* Is it possible to measure health -related quality of life?
* What impact does the novel radiotherapy approach have on: patient's quality of life, control of the brain metastasis (control of the lesion) and steroid use?

Participants will:

* Receive 5 doses of radiotherapy
* Complete weekly quality of life (EQ-5D) assessments and medication (steroid) diaries (via telephone/ postal) until 12 weeks post enrolment
* Be reviewed in clinic with up-to-date MRI scans at 8, 12 and 24 weeks post-enrolment
* Complete a more detailed HRQoL panel of assessments will be assessed at baseline, 8 weeks, 12 weeks and 24 weeks post enrolment.

DETAILED DESCRIPTION:
Brain metastases from breast cancer are a common, and devastating, complication with survival times of 3 - 5 months from diagnosis.

The main treatment approaches to brain metastases are surgery, stereotactic radiosurgery (SRS), and whole brain radiotherapy. However, it is known that most patients with brain metastases receive either whole-brain radiotherapy (WBRT) or no treatment, with relatively low rates of surgery and SRS. Since the commonest treatment in those who do have treatment is WBRT, the local team have developed an approach that is believed to be (possibly) more effective than WBRT. The objective is to evaluate this approach in patients who are not suitable to receive more aggressive treatment and who would otherwise receive WBRT. The local approach involves using a modern radiotherapy planning approach, combined with careful, intra-metastasis dose escalation (Dose Escalated internal PTV (DE-iPTV)) to deliver a higher dose to tumour, while delivering less dose to the brain. The combination of less dose to normal structures and more dose to the lesion will hopefully improve Health-related Quality of Life (HRQoL).

The aim of this study is to demonstrate the feasibility of delivering complex radiotherapy, dose escalated internal PTV (DE-iPTV), and measuring quality of life at 8 weeks post-enrolment for patients with brain metastases from breast cancer who would otherwise receive WBRT. An exploratory blood-based biomarker sample collection and analysis will be completed. Furthermore, linked national cancer data will be used to measure the number of patients currently offered WBRT, including survival costs and hospital admissions, and thus provide a baseline to estimate the impact of this novel approach.

ELIGIBILITY:
Inclusion Criteria

1. Written (signed and dated) informed consent and be capable of co-operating with treatment and follow-up
2. Adult (aged 16+) patients, resident in the United Kingdom.
3. Histologically confirmed primary breast cancer with brain metastases on MRI imaging
4. The treating oncologist considers whole-brain radiotherapy to be the most suitable treatment outside of the trial.
5. Eastern Cooperative Oncology Group Performance status 0, 1 or 2
6. Able to respond to question about their quality of life, symptoms, and side effects remotely (via telephone assessments
7. Life expectancy from extra-cranial disease >3 months

Exclusion Criteria

1. Leptomeningeal disease
2. "Miliary" pattern of metastases: patients with over 15 metastases are excluded (clinician-based assessment)
3. Cystic metastases
4. Previous whole or partial brain radiotherapy (previous surgery or SRS is acceptable)
5. Plan for hippocampal-sparing whole brain radiotherapy.
6. Unable to give informed consent.
7. Prognosis less than 3 months
8. Pregnant or nursing women
9. Unable to complete a brain MRI and/or known allergy to gadolinium.

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-01-06 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of delivering DE-iPTV and measuring health related quality of life questionnaire in patients with brain metastases from breast cancer to whom their treating clinician would normally offer whole brain radiotherapy | 8 weeks post-enrolment
  Completion of radiotherapy and completion of EuroQol- 5 Dimension (EQ-5D-5L) questionnaire

SECONDARY OUTCOMES:
Lesional Response | 8 weeks
  Lesional response and intracranial progression measured using RANO-BM criteria
Intracranial progression | 3 months
  Intracranial progression based on RANO-BM
Intracranial progression | 6 months
  Intracranial progression based on RANO-BM
Treatments | Within 6 months of enrolment
  Use of further brain-directed therapies (reported by clinician)
Central Nervous System (CNS) Failures | Within 6 months of enrolment
  Time to CNS failure (either lesional progression or developing a new lesion as per RANO-BM)
Neurological toxicities | Within 6 months of enrolment
  Acute and late neurological/ CNS toxicity as assessed using CTCAE v5
Health Related Quality of Life | Within 6 months of enrolment
  HRQoL over time (participants reported outcomes for descriptive analysis)
Time to deterioration in quality of life | Within 6 months of enrolment
  Time to deterioration in Health Related Quality of Life - measured as time to first time there is a minimum clinically significant change in EuroQol- 5 Dimension (EQ-5D-5L)
Symptom Burden | Within 6 months of enrolment
  Symptom burden assessed by collection of clinician-recorded toxicities
Steroid usage | Within 6 months of enrolment
  Use of corticosteroids over time, assessed through clinician reports and patient diaries
Quality-Adjusted Life Year | Within 6 months of enrolment
  Quality-Adjusted Life Year
Overall survival | End of study
  Overall survival

OTHER OUTCOMES:
Changes in blood-based biomarkers | 8 weeks
  Change between baseline and week 8 levels of Circulating Tumour DNA (ctDNA) and S100
Imaging Changes | Up to 6 months post enrolment
  MRI-based response (as per RANO-BM and serial volumetric measurements)
Radiation Necrosis | Up to 6 months post enrolment
  Radiation necrosis based on radiologist report

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen J, Sinclair G, Rozati H, Hill L, Pakzad-Shahabi L, Wang J, Calvez KL, Paddick I, Williams M. Improving on whole-brain radiotherapy in patients with large brain metastases: A planning study to support the AROMA clinical trial. Radiother Oncol. 2022 May;170:176-183. doi: 10.1016/j.radonc.2022.02.011. Epub 2022 Feb 17. PMID 35182688
- See also: Related Info — https://www.computationaloncology.net/aroma